CLINICAL TRIAL: NCT04196400
Title: Prospective Comparative Trial to Assess the Role of Local Long Acting Steroid Injection After Hypospadias Surgery in Decreasing Complications and Preserving Better Cosmesis
Brief Title: The Role of Local Long Acting Corticosteroid Injection in Hypospadias Surgery.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abozamel, Doctor Lecturer in Urology department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Hypospadias-101
Record Dates: First submitted 2019-12-09; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Hypospadias
Keywords: hypospadias, edema, failure, fistula, steroids
MeSH Terms: conditions — Hypospadias; Edema; Fistula

STUDY DESIGN:
Intervention Model Description: comparative prospective clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Steroid injection (Active Comparator): Steroid (betamethasone) 2 ml is injected subcutaneously after finishing the operation at the repair site.
  Interventions: Drug: steroid betamethasone
- Control Group (No Intervention)

INTERVENTIONS:
Drug: steroid betamethasone — The steroid is injected using insulin needle in the subcutaneous tissue after finishing the repair
  Arms: Steroid injection

SUMMARY:
Post-operative tissue oedema is one of the main causes of failure of hypospadias repair. Severe oedema may disrupt the suture line, invite infection and result in repair failure. Thus, we suggested that local injection of corticosteroids in just below coronal sulcus into dartos and buck's fascia may limit this oedema thus improving the outcome of hypospadias repair.

DETAILED DESCRIPTION:
This is a prospective comparative trial : comparing the use of local steroids injection to reduce tissue edema after hypospadias and to preserve the final cosmesis after tissue repair.

The patients will be divided into 2 groups(each group 20 patients): one group will be injected steroids just after hypospadias surgery while the other will not.

The short and long term outcomes between both groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Hypospadias Patient
* Recurrent Cases
* 6 months or more
* Distal, and mid penile hypospadias

Exclusion Criteria:

* None

Min Age: 6 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Failure rate | 2 weeks

SECONDARY OUTCOMES:
incidence of Tissue edema | 3 days, 5 days, 10 days, 2 weeks
Infection Rate | 3 days, 5 days, 10 days, 2 weeks
Fistula rate | 2 weeks
Final cosmesis | 3 days, 5 days, 10 days, 2 weeks
  The shape of the glans penis and surrounding tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo Univeristy Hospital, Cairo, Egypt